CLINICAL TRIAL: NCT06887348
Title: Long-term Safety Outcomes in Patients Treated With Replimune Oncolytic Immunotherapy Products
Brief Title: A Study to Assess the Long-term Safety Outcomes in Patients Previously Treated With RP1, RP2, or RP3
Acronym: RPx
Status: Recruiting | Type: Observational
Sponsor: Replimune Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RPL-123-01
Expanded Access: NCT06590480 (No longer available)
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Melanoma; Metastatic Melanoma; Advanced Solid Tumor; Hepatocellular Carcinoma
Keywords: Advanced solid tumors; Immunotherapy; Immuno-oncology; Oncolytic virus; Oncolytic immuno-gene therapy; Hepatocellular Carcinoma; Cutaneous Melanoma; Anti-PD1 failed; Non-melanoma Skin Cancer; Melanoma (skin)
MeSH Terms: conditions — Melanoma; Carcinoma, Hepatocellular | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients who received at least 1 dose of an RPx [RP1, RP2, RP3]: This is an observational study and there will be no clinical interventions.
  Interventions: Other: Observational study with no interventions

INTERVENTIONS:
Other: Observational study with no interventions — This is an observational study and there will be no clinical interventions.
  Other Names: Observational Study

SUMMARY:
This is a noninterventional, observational, long-term follow-up (LTFU) study. Patients in this study will be followed for 5 years from enrollment on this study to assess potential delayed risks of RPx products. Eligible participants for this LTFU study include patients who received at least 1 dose of an RPx product under the interventional parent study. Patients will be rolled over into this LTFU study after completion of the Replimune-sponsored parent study (ie, either completion of the LTFU in the parent study or withdrawal from the parent study). All patients in ongoing RPx studies will be asked to participate in this LTFU study so that the Sponsor can evaluate potential delayed risks.

DETAILED DESCRIPTION:
Long-term outcomes include detection of delayed adverse event(s) for any new malignancy(ies), new incidence or exacerbation of a pre-existing neurologic disorder, rheumatologic or other autoimmune disorder, hematologic disorder, new incidence of infection related to RPx product and new incidence of herpetic-like infection. Patients with a suspected herpetic infection will be asked to provide a sample of the area of the suspected infection (using a swab), and also may be asked to provide additional biological samples (eg, a blood or urine sample to determine presence of RPx.) No study interventions will be administered in this observational study. Patients will be contacted by telephone every 3 months (Q3M) for 5 years from enrollment on this study. Participant visits may occur in person, over the phone, by video conference, or other technology.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for inclusion in the study only if they meet all of the following criteria:

1. Patient has received at least 1 dose of an RPx product and has completed or discontinued participation in the parent study.
2. Patient or patient's legal guardian has provided signed informed consent (or assent) as , which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

Patients are excluded from the study if the following criterion applies:

1. Cannot comply with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are eligible for inclusion in the study only if they meet all of the inclusion criteria.
  Deviations from the entry criteria that would be considered a protocol waiver or exemption are not permitted.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the long-term safety of patients treated with an RPx product | Every 3 months (Q3M) (± 30 days) for 5 years from enrollment on this study to assess potential delayed risks
Identify any delayed adverse event(s) related to treatment with an RPx product | Every 3 months (Q3M) (± 30 days) for 5 years from enrollment on this study to assess potential delayed risks
Identify systemic HSV-1 infection related to treatment with an RPx product | Every 3 months (Q3M) (± 30 days) for 5 years from enrollment on this study to assess potential delayed risks

CONTACTS AND LOCATIONS:
Locations (2):
- UC San Diego Moores Cancer Center, La Jolla, California, United States
- Tasman Oncology Research, Southport, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No